CLINICAL TRIAL: NCT04011410
Title: Phase 2 Study of Hydroxychloroquine to Increase Tumor Suppressor PAR-4 Levels in Oligometastatic Prostate Cancer
Brief Title: Hydroxychloroquine to Increase Tumor Suppressor PAR-4 Levels in Oligometastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Patrick Hensley (Other)
Responsible Party: Sponsor-Investigator, Patrick Hensley, Assistant Professor, Dept of Urology, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 50146 - MCC-19-GU-72
Record Dates: First submitted 2019-07-01; First posted 2019-07-08 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer Recurrent
Keywords: Prostate Cancer; Oligometastatic Prostate Cancer; Limited Metastatic Disease; Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Single arm, non-blinded, open label clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Hydroxychloroquine (Experimental): Hydroxychloroquine (HCQ)
  DOSAGE FORM: 200 mg tablet, oral route
  DOSAGE: 200 mg BID by mouth, for a total daily dose of 400 mg
  FREQUENCY: HCQ is taken twice daily (morning and night) with food.
  DURACTION OF HCQ: 90-days
  Interventions: Drug: Hydroxychloroquine Sulfate 200Mg Tab

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate 200Mg Tab — Twice daily for 90-days, administered two weeks prior to radiation/surgery of oligometastatic lesions
  Other Names: Hydroxychloroquine; plaquenil; plaquenil sulfate; quineprox

SUMMARY:
Treatment of recurrent oligometastatic prostate cancer may be enhanced by the addition of Hydroxychloroquine to the current treatment regimens. Potential benefits of Hydroxychloroquine include delayed disease progression and delayed initiation of androgen deprivation therapy (ADT), thus lessening morbidity, distressing side effects, and improving functioning and quality of life in men with recurrent prostate cancer.

Building on prior research at Markey, patients recently diagnosed with recurrent oligometastatic prostate cancer will be approached about participating in this study. Per standard of care, these patients undergo either surgery or radiation, in addition participants of this clinical trial will also receive Hydroxychloroquine (400 mg per day, oral medication) for 3 months.

It is expected that a participant will exhibit a 50% increase of tumor suppressor PAR-4, as well as few, if any, negative side effects from Hydroxychloroquine.

DETAILED DESCRIPTION:
This investigator-initiated clinical trial (IIT) builds on and extends research on autophagy in prostate cancer with PAR-4 and HCQ conducted by a transdisciplinary investigative team, and is sponsored by funding from Markey Cancer Center.

Prostate cancer is the most common cancer in men and the 2nd most common cause of cancer death in men. Secondary to the greying of the U.S. population and increasing life expectancy, metastatic prostate cancer (mPCa) rates are increasing. Androgen deprivation therapy (ADT) has been the primary treatment for metastatic prostate cancer. The survival benefit of ADT is juxtaposed against significant adverse effects including cardiovascular morbidity, skeletal fractures, diabetes, sexual dysfunction, and a decrease in cognitive function. Recent studies have indicated a potential benefit to treatment of metastatic lesions in men with limited metastatic disease and have identified a potential delay in initiation of ADT in men whose limited metastatic lesions were treated with stereotactic radiotherapy. Prostate apoptosis response-4 (PAR-4) is a tumor suppressor protein that facilitates apoptosis in numerous types of cancer cells. Hydroxychloroquine (HCQ) has been found to induce PAR-4 expression and subsequently promote apoptosis of cancer cells and inhibit metastatic progression. HCQ has also been reported to both inhibit and enhance immune responses via changes in Th1, Th2, Th17 and Treg subsets and reduce inflammatory markers. It also acidifies lysosomes which potentially inhibits antigen presentation by antigen-presenting cells, and can be measured with LysoSensor Yellow/Blue DND-160 by flow cytometry and induces autophagy which can be detected by measuring up-regulation of the microtubule associated protein LC3B. Treatment of oligometastatic prostate cancer may be enhanced by the addition of Hydroxychloroquine to either surgical resection or radiation treatment of metastatic lesions. Potential benefits of Hydroxychloroquine include delayed disease progression and delayed initiation of ADT, lessening morbidity and increasing quality of life in men with oligometastatic prostate cancer.

A single-arm, open-label phase II trial will be conducted in a population of men with recurrent oligometastatic prostate cancer following primary treatment of localized disease. The oligometastatic sites will be treated with either surgical resection or stereotactic radiation per standard of care, in addition to 400 mg of Hydroxychloroquine per day for a period of 3 months.

Sample Size:

Based on an ongoing Phase I trial of HCQ, the proportion of patients who will exhibit a 50% induction in PAR-4 from baseline levels is equal to 0.50, compared to a null hypothesis of 0.20. A sample of 18 patients will provide 84% power to detect this hypothesized difference in proportion based on a two-sided test with 5% significance level. Prior studies at Markey Cancer Center in this population have demonstrated an attrition rate of less than a 10%. Thus, a total of 20 patients will be enrolled into the study.

Specific and Secondary Aims:

The primary objective is to assess the rate of attainment of a 50% increase in tumor suppressor PAR-4 levels from baseline in patients treated with 3-months of hydroxychloroquine (HCQ), in combination with radiation or surgery for recurrent, oligometastatic prostate cancer.

Secondary aims of the trial include assessment of: median progression-free survival; 1- and 3-year ADT-free survival; treatment toxicity and quality of life.

Correlative studies of the trial comprise assessment of immunological effect of Hydroxychloroquine by analyzing peripheral blood mononuclear cells (PBMC's).

Statistical Analytic Plan:

Descriptive statistics will be calculated to summarize PAR-4 levels at each time point of follow-up. Percent change from baseline compared to each follow-up time point will likewise be calculated. The proportion of patients who exhibit a 50% induction in PAR-4 compared to baseline within the 3-month therapy period will be calculated and a one-sample test for proportion will be performed. Secondary analyses of the primary endpoint will also be performed. Continuous changes in PAR-4 levels will also be assessed using paired t-test or nonparametric analog. Linear mixed models will be employed to analyzed repeatedly measured levels of PAR-4 and association with clinical parameters as well as PSA levels.

* Other secondary analyses will include summary of the PAR-4 induction profile over the 3-month treatment period and after end of therapy period. PSA levels will be assessed and PSA doubling time will be calculated. Association of PSA levels with PAR-4 levels will be determined using Spearman or Pearson's correlation coefficient. Quality of life as measured by the EORTC QLQ-C30 supplemented with QLQ-PR25 will be evaluated and descriptive statistics of QOL scores will be calculated. Association of QOL with PAR-4, PSA and other clinical endpoints will be determined in an exploratory manner using correlations and survival analysis models.
* All participants who received HCQ will be included in the safety analysis. Frequency and incidence tables of toxicity and AEs will be generated.
* Immune outcome endpoints including markers of immune function/activation and systemic inflammation will be summarized at each time point of follow-up. Linear mixed models will be utilized to model these repeatedly measured immune endpoints to determine changes over time. Associations between markers and PAR-4 levels will be assessed via calculation and comparison of correlation coefficients. Data processing, data analysis pipelines and bioinformatics methods for NGS data will be employed in collaboration with MCC Shared Resource Facilities. False discovery rate (FDR) q values will be calculated for multiple comparison adjustment, with threshold significance set to 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer that has recurred
* Three or fewer synchronous metastatic lesions (on imaging) with no evidence of residual local disease
* ECOG performance status 0 - 2
* Approval by screening eye exam (disqualifying baseline conditions listed below)
* Ability to provide informed consent

Exclusion Criteria:

* Receipt of hydroxychloroquine (HCQ) within the past 6 months
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to HCQ
* Use of contraindicated medications,
* Macular degeneration
* Cataracts
* Severe baseline visual impairment, retinopathy or visual field changes
* Presence of only one functional eye
* Prior treatment with ADT including:
* Previous history of radiation or surgery to a metastatic site
* Serum testosterone less than 50 ng/ml
* History of orchiectomy
* History of pathologic fracture or spinal cord compression
* Brain or CNS metastases
* History of G-6-PD (glucose-6-phosphate dehydrogenase) deficiency
* Uncontrolled intercurrent illness
* Psychiatric illness and/or social situations that would limit compliance with study requirements.
* Patients taking other investigational agents

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Hensley, MD, Principal Investigator — University of Kentucky; Peng Wang, MD, Principal Investigator — University of Kentucky
Locations (1):
- Markey Cancer Center - University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication detailing the primary endpoint
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after publication

REFERENCES:
- [Background] Tosoian JJ, Gorin MA, Ross AE, Pienta KJ, Tran PT, Schaeffer EM. Oligometastatic prostate cancer: definitions, clinical outcomes, and treatment considerations. Nat Rev Urol. 2017 Jan;14(1):15-25. doi: 10.1038/nrurol.2016.175. Epub 2016 Oct 11. PMID 27725639
- [Background] Taylor LG, Canfield SE, Du XL. Review of major adverse effects of androgen-deprivation therapy in men with prostate cancer. Cancer. 2009 Jun 1;115(11):2388-99. doi: 10.1002/cncr.24283. PMID 19399748
- [Background] Burikhanov R, Shrestha-Bhattarai T, Hebbar N, Qiu S, Zhao Y, Zambetti GP, Rangnekar VM. Paracrine apoptotic effect of p53 mediated by tumor suppressor Par-4. Cell Rep. 2014 Jan 30;6(2):271-7. doi: 10.1016/j.celrep.2013.12.020. Epub 2014 Jan 9. PMID 24412360
- [Background] Hebbar N, Wang C, Rangnekar VM. Mechanisms of apoptosis by the tumor suppressor Par-4. J Cell Physiol. 2012 Dec;227(12):3715-21. doi: 10.1002/jcp.24098. PMID 22552839
- [Background] Kimura T, Takabatake Y, Takahashi A, Isaka Y. Chloroquine in cancer therapy: a double-edged sword of autophagy. Cancer Res. 2013 Jan 1;73(1):3-7. doi: 10.1158/0008-5472.CAN-12-2464. PMID 23288916
- [Background] Ratikan JA, Sayre JW, Schaue D. Chloroquine engages the immune system to eradicate irradiated breast tumors in mice. Int J Radiat Oncol Biol Phys. 2013 Nov 15;87(4):761-8. doi: 10.1016/j.ijrobp.2013.07.024. PMID 24138918
- [Background] Burikhanov R, Hebbar N, Noothi SK, Shukla N, Sledziona J, Araujo N, Kudrimoti M, Wang QJ, Watt DS, Welch DR, Maranchie J, Harada A, Rangnekar VM. Chloroquine-Inducible Par-4 Secretion Is Essential for Tumor Cell Apoptosis and Inhibition of Metastasis. Cell Rep. 2017 Jan 10;18(2):508-519. doi: 10.1016/j.celrep.2016.12.051. PMID 28076793
- [Background] Wang P, Burikhanov R, Jayswal R, Weiss HL, Arnold SM, Villano JL, Rangnekar VM. Neoadjuvant administration of hydroxychloroquine in a phase 1 clinical trial induced plasma Par-4 levels and apoptosis in diverse tumors. Genes Cancer. 2018 May;9(5-6):190-197. doi: 10.18632/genesandcancer.181. PMID 30603055

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydroxychloroquine: Hydroxychloroquine (HCQ)
  DOSAGE FORM: 200 mg tablet, oral route
  DOSAGE: 200 mg BID by mouth, for a total daily dose of 400 mg
  FREQUENCY: HCQ is taken twice daily (morning and night) with food.
  DURACTION OF HCQ: 90-days
  Hydroxychloroquine Sulfate 200Mg Tab: Twice daily for 90-days, administered two weeks prior to radiation/surgery of oligometastatic lesions
Period: Overall Study
Arm/Group | Hydroxychloroquine
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Hydroxychloroquine
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: years] | 69 [55 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Participants With Greater Than or Equal to 50% Induction in Serum PAR4 Levels
Description: Number of participants that attained greater than or equal to 50% induction over baseline of PAR-4 levels as measured via serum or plasma blood sample
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine
Number analyzed (Participants) | 19
Participants | 11

2. Secondary Outcome: Change in Serum Prostate Specific Antigen (PSA) Levels
Description: Doubling time of serum PSA levels
Time Frame: 5 timepoints: baseline, 30-, & 90-days post-HCQ initiation; and at 6- and 12-mos follow-up
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Hydroxychloroquine
Number analyzed (Participants) | 19
ng/ml
  Baseline | 8.60 (8.373)
  30 days | 10.91 (10.875)
  90 days | 14.46 (23.281)
  6 months | 7.54 (12.190)
  12 months | 0.38 (0.794)

3. Secondary Outcome: Number of Participants With Progression-Free Survival
Description: Assessed via imaging per standard of care using Response Evaluation Criteria in Solid Tumours (RECIST) scoring criteria
Time Frame: 1 year progression free survival
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine
Number analyzed (Participants) | 19
Participants | 6

4. Secondary Outcome: Number of Participants With Androgen Deprivation Therapy (ADT)-Free Survival
Description: ADT-free Survival is defined as the time between study enrollment until the start of ADT or death
Time Frame: 1 year ADT free survival
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxychloroquine
Number analyzed (Participants) | 19
Participants | 8

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from study enrollment up to 12 months after study initiation.
Arm/Group | Hydroxychloroquine
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 9/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=19)
Gastrointestinal distress (Gastrointestinal disorders) | 9 (9)
Generalized distress (fatigue/pain) (General disorders) | 5 (5)
Metabolic disturbance (Metabolism and nutrition disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT04011410/Prot_SAP_000.pdf